CLINICAL TRIAL: NCT02680795
Title: Open-label, Nonrandomized, Phase 1 Study Evaluating Safety and Pharmacokinetics of Belinostat in Patients With Relapsed/Refractory Solid Tumors or Hematological Malignancies in Wild-Type, Heterozygous, and Homozygous UGT1A1*28 Genotypes
Brief Title: Establish the PK of Belinostat in Patients With Wild-type, Heterozygous, and Homozygous UGT1A1*28 Genotypes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Axis Clinicals Limited (Industry); Axis Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-BEL-106
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors; Hematological Malignancies
Keywords: UGT1A1*28; Belinostat; beleodaq; wild type genotypes; heterozygous genotypes; homozygous genotypes
MeSH Terms: conditions — Hematologic Neoplasms | interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wild Type UGT1A1 (Experimental): Cohort A: Open for Enrollment Wild Type UGT1A1, Belinostat IV
  Interventions: Drug: Belinostat IV
- Heterozygous UGT1A1*28 (Experimental): Cohort B: Closed For Enrollment Heterozygous UGT1A1, Belinostat IV
  Interventions: Drug: Belinostat IV
- Homozygous UGT1A1*28 (Experimental): Cohort C: Open For Enrollment Homozygous UGT1A1, Belinostat IV
  Interventions: Drug: Belinostat IV

INTERVENTIONS:
Drug: Belinostat IV — Cohort A:
  Belinostat 1000mg will be administered once daily on days 1 through 5 of one 21-day cycle via 30-minute IV infusion.
  Cohort B:
  Belinostat 1000mg will be administered once daily on days 1 through 5 of one 21-day cycle via 30-minute IV infusion.
  Cohort C:
  Belinostat 750mg will be administered once daily on days 1 through 5 of one 21-day cycle via 30-minute IV infusion.
  Other Names: Beleodaq

SUMMARY:
This is a Phase 1, open-label, nonrandomized study to determine the PK profiles of belinostat in patients with relapsed/refractory solid tumors or hematological malignancies who have heterozygous and homozygous UGT1A1*28 genotypes and wild-type UGT1A1 gene. Enrolled patients will be assigned to 1 of 3 cohorts (A, B, or C) based on their UGT1A1 genotype

DETAILED DESCRIPTION:
This is a Phase 1, open-label, nonrandomized study to determine the PK profiles of belinostat in patients with relapsed/refractory solid tumors or hematological malignancies who have heterozygous and homozygous UGT1A1*28 genotypes and wild-type UGT1A1 gene. Enrolled patients will be assigned to 1 of 3 cohorts (A, B, or C) based on their UGT1A1 genotype

Enrollment into all cohorts will occur simultaneously rather than sequentially. Belinostat will be administered via a 30-minute infusion once daily from Day 1 to Day 5 of one 21-day cycle. Clinical safety will be monitored in each patient. Blood samples for PK analysis will be collected from Day 1 to Day 3, and urine samples for PK analysis will be collected from Day 1 to Day 4.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is diagnosed with advanced solid tumors or advanced hematological malignancy that is relapsed/refractory, for which no standard salvage therapy exists.
2. Patient must have received at least 1 prior systemic therapy for the current malignancy and has recovered from any toxicity of the prior therapy at screening.
3. Patient has adequate hematological and hepatic functions.

Exclusion Criteria:

1. Patient is taking UGT1A1 inhibitors (eg, atazanavir, gemfibrozil, indinavir, ketoconazole, sorafenib) at screening.
2. Patient has HBV or HCV
3. Patient has a known HIV positive diagnosis.
4. Patient has congestive heart failure Class III/IV
5. Patient has had previous exposure to belinostat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Plasma and urine concentrations of belinostat will be measured | 26 Weeks
  PK will be measured for area under the time-concentration curve (AUC), steady state volume of distribution (Vdss),PK will be measured for total body clearance (CLtot),PK will be measured for fraction excreted unchanged (fe), PK will be measured for renal clearance (CLren), PK will be measured for non-renal clearance (CLnonren), PK will be measured for peak concentration (Cmax),and half-life (t1/2)

SECONDARY OUTCOMES:
Assess overall incidence of treatment emergent adverse events (TEAEs) using CTCAE version 4.03 | 26 Weeks
  Assess Safety of belinostat in patients with wild type, heterozygous, and homozygousUGT1A1*28 genotypes
Assess any adverse events (AEs) (changes in physical exam or laboratory findings related to study medication dosing | 26 Weeks
  Assess Safety of belinostat in patients with wild type, heterozygous, and homozygousUGT1A1*28 genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Khan, MD, Study Director — Acrotech Biopharma Inc.
Locations (3):
- United States (3):
  - John Wayne Cancer Institute @ Providence Saint John's Health Center, Santa Monica, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Gabrail Cancer Center Research, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No